CLINICAL TRIAL: NCT02592109
Title: Effect of Enhanced Counseling Using Complementary Feeding Recommendation Based on Linear Programming on Nutritional Status, Omega-3 Fatty Acid, Malondialdehyde, and Alpha-Tocopherol in Children With Risk of Overweight in East Jakarta
Brief Title: Effect of Enhanced Counseling Using Complementary Feeding Recommendation Based on Linear Programming on Nutritional Status,Omega-3 Fatty Acids, Malondialdehyde, and Alpha-Tocopherol in Overweight Children in East Jakarta
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Danone Institute International (Other)
Responsible Party: Principal Investigator, Inge Permadhi, Dr. dr. MS SpGK, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IPermadhi
Record Dates: First submitted 2015-10-29; First posted 2015-10-30 (Estimated); Last update posted 2016-06-22 (Estimated); Status verified 2016-06

CONDITIONS: Complementary Feeding Recommendation; Linear Programming,; Nutritional Status; Omega-3 Fatty Acids; Malondialdehyde; Alpha-Tocopherol; Overweight
Keywords: Complementary Feeding Recommendation; Linear Programming; Nutritional Status; Omega-3 Fatty Acids; Malondialdehyde; alpha-Tocopherol
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Counseling using CFR based on LP (Experimental): The counseling will be done by individual face-to-face communications. The intervention's arm will get a counseling with an additional of 7-day cycle with adequate n-3 and optimal n-3/6 ratio for complementary feeding menu obtained from linear programming formulation.
  The counseling consisted of nutritional status in children aged 12-23 months and how to determine the nutritional status; the principle of balanced diet; definition, function, and source of omega-3; example of menu that contains adequate omega-3. The duration of counseling is approximately 30 minutes, once a week for ten weeks. The mother or caregiver will also receive daily menu for seven days that should be followed during the intervention. The daily menu comprised of 3 main meals and 2 snacks.
  Interventions: Behavioral: Enhanced Counseling using CFR based on Linear Programming
- General CFR Counseling (Active Comparator): The control's arm will get general counseling combining balance diet and IYCF principal, which already been used by Ministry of Health, with additional of 7-day cycle menu guidance modified from existing or available menu which can be downloaded for public on Ministry of Health official website.
  The counseling consisted of nutritional status in children aged 12-23 months and how to determine the nutritional status; the principle of balanced diet based on Ministry of Health's Recommendation, and example of balanced diet menu. The duration of counseling is approximately 30 minutes, once a week for ten weeks. The mother or caregiver will also receive daily menu for seven days that should be followed during the intervention. The daily menu comprised of 3 main meals and 2 snacks.
  Interventions: Behavioral: Enhanced Counseling using CFR based on Linear Programming

INTERVENTIONS:
Behavioral: Enhanced Counseling using CFR based on Linear Programming

SUMMARY:
The epidemic of pediatric obesity has become a public health burden in both developed and developing countries, due to its serious health consequences, including an increased risk of type 2 Diabetes Mellitus and heart disease. Currently, dietary and exercise changes are still the center of preventive and treatment measures of obesity. Recently, the omega-3 group, one of the groups of polyunsaturated fatty acids (PUFAs), has been associated with many positive effects leading to the improvement of many diseases related to obesity. Nevertheless, the consumption of this essential nutrient requires certain ration to optimize its favorable result. Although previous studies have examined the efficacy of dietary counseling approach as treatment for obesity, none of them as explicitly explore the use of linear programming to create a tailored diet containing high omega-3 fatty acid food as a part of dietary counseling in obesity management program among children. Thus, this study is intended to contribute the clinical evidence regarding this area of knowledge, specifically the effects of enhanced counseling containing complementary feeding recommendation on nutritional status, omega-3 fatty acid, malondialdehyde, and alpha Tocopherol among children with risk of overweight aged 12 -23 months in East Jakarta.

DETAILED DESCRIPTION:
Randomized-Controlled-Trial with two arms of intervention:

1. Control group: receive standard counseling with general existing menu recommendation
2. Intervention group: receive enhanced counseling (additional information on omega-3 fatty acids) with population-based menu ganerated from linear programming (LP)

There is a protocol on stratified block randomization. 2 blocks, stratified by: area, age, BMI-for-age status.

Total sample size for analysis:

Overall: 20 control - 18 intervention Blood sample: 18 control - 14 intervention

ELIGIBILITY:
Inclusion Criteria:

* aged 12-23 months old at first counseling
* body mass index more than +1 standard deviation in WHO Z-score
* parent agree to participate in the study by signing informed consent

Exclusion Criteria:

* Children with congenital disease and serious diseases
* Children with parent/caregiver who is illiterate
* Children with parent/caregiver who had communication disability

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Nutritional status | 10 weeks
  Body weight and body height will be used to calculate body mass index

SECONDARY OUTCOMES:
Omega-3 Fatty Acid in plasma | 10 weeks
Malondialdehyde plasma | 10 weeks
alpha-Tocopherol plasma | 10 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Posyandu di Kelurahan Pisangan Timur, Cipinang, Kayuputih, Rawamangun, Jakarta, DKI Jakarta, Indonesia